CLINICAL TRIAL: NCT00006251
Title: Induction of Mixed Hematopoietic Chimerism in Patients Using Fludarabine, Low Dose TBI, PBSC Infusion and Post-Transplant Immunosuppression With Cyclosporine and Mycophenolate Mofetil
Brief Title: Fludarabine Phosphate, Low-Dose Total-Body Irradiation, and Donor Stem Cell Transplant Followed by Cyclosporine, Mycophenolate Mofetil, Donor Lymphocyte Infusion in Treating Patients With Hematopoietic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1533.00; NCI-2013-01634 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1533.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P01CA078902 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2000-09-11; First posted 2004-06-09 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Acute Undifferentiated Leukemia; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Childhood Burkitt Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Myelomonocytic Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Juvenile Myelomonocytic Leukemia; Mast Cell Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Myeloid/NK-cell Acute Leukemia; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Primary Systemic Amyloidosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Renal Cell Cancer; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage II Multiple Myeloma; Stage III Multiple Myeloma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myelomonocytic, Chronic; Intraocular Lymphoma; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Immunoglobulin Light-chain Amyloidosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Renal Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Whole-Body Irradiation; fludarabine phosphate; Cyclosporine; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (fludarabine phosphate, TBI, PBSC transplant, DLI) (Experimental): CONDITIONING REGIMEN : Patients receive fludarabine phosphate IV on days - 4 to -2 and undergo low-dose TBI on day 0. (Note: Patients who have had an autologous transplant within 90 days prior to day 0 will not receive fludarabine phosphate.)
  PBSC INFUSION: Patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID on days -3 to 35 with a taper to day 56. Patients receive mycophenolate mofetil PO BID on days 0-27.
  POST TRANSPLANT DLI: Patients with stable mixed chimerism on day 56, and without evidence of GVHD, undergo DLI IV over 30 minutes on day 65. Patients without a complete response, full donor chimerism, and GVHD after 2 months undergo further DLI at higher cell numbers. Up to 6 DLIs may be given 65 days apart.
  Interventions: Radiation: total-body irradiation; Drug: fludarabine phosphate; Drug: cyclosporine; Drug: mycophenolate mofetil; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Biological: donor lymphocytes; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cyclosporine — Given PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSC transplant
Biological: donor lymphocytes — Undergo DLI
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies fludarabine phosphate, low-dose total-body irradiation, and donor stem cell transplant followed by cyclosporine, mycophenolate mofetil, and donor lymphocyte infusion in treating patients with hematopoietic cancer. Giving low doses of chemotherapy, such as fludarabine phosphate, and total body irradiation (TBI) before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also keep the patient's immune response from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the risk of graft rejection associated with the addition of fludarabine (fludarabine phosphate) to a non-myeloablative conditioning regimen for patients with malignant diseases treatable by allogeneic stem cell transplantation and compare this rate to that observed among patients previously treated without fludarabine.

II. To estimate the rate of grade acute II/IV graft-vs-host disease (GVHD) and chronic GVHD in patients treated with low-dose total-body irradiation (TBI), fludarabine, peripheral blood stem cell (PBSC) infusion and immunosuppression with cyclosporine and mycophenolate mofetil.

OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days - 4 to -2 and undergo low-dose TBI on day 0. (Note: Patients who have had an autologous transplant within 90 days prior to day 0 will not receive fludarabine phosphate.)

PBSC INFUSION: Patients undergo allogeneic PBSC transplant on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) twice daily (BID) on days -3 to 35 with a taper to day 56. Patients receive mycophenolate mofetil PO BID on days 0-27.

POST TRANSPLANT DONOR LYMPHOCYTE INFUSION (DLI): Patients with stable mixed chimerism on day 56, and without evidence of GVHD, undergo DLI IV over 30 minutes on day 65. Patients without a complete response, full donor chimerism, and GVHD after 2 months undergo further DLI at higher cell numbers. Up to 6 DLIs may be given 65 days apart.

After completion of study treatment, patients are followed up at 4, 6, 12, 18 and 24 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 49 years and < 75 years with non-Hodgkin lymphoma (NHL), chronic lymphocytic leukemia (CLL) and multiple myeloma who are not eligible for a curative autologous transplantation or who have failed prior autologous transplantation; patients with NHL and CLL must have failed prior therapy with an alkylating agent and/or fludarabine, or be at high risk of relapse; patients with multiple myeloma must have stage II or III disease and received prior chemotherapy
* Patients < 50 years of age with NHL, CLL or multiple myeloma at high risk of regimen related toxicity through prior autologous transplant or through pre-existing medical conditions
* Patients < 75 years of age with other malignant diseases treatable by allogeneic bone marrow transplant (BMT) whom through pre-existing chronic disease affecting kidneys, liver, lungs, and heart are considered to be at high risk for regimen related toxicity using standard high dose regimens; the following diseases are the likely candidates:

  * Myelodysplastic syndromes
  * Myeloproliferative syndromes
  * Acute Leukemia with < 10% blasts
  * Amyloidosis
  * Hodgkin's disease
  * Renal cell carcinoma
* Patients with other malignancies declining standard allografts may be approved for transplant following presentation and approval by the Fred Hutchinson Cancer Research Center (FHCRC) chimerism group
* DONOR:

  * Human leukocyte antigen (HLA) genotypically or phenotypically identical related donor
  * Donor must consent to granulocyte colony-stimulating factor (G-CSF) administration and leukopheresis
  * Donor must have adequate veins for leukopheresis or agree to placement of central venous catheter (femoral, subclavian)
  * Age < 75 years

Exclusion Criteria:

* Eligible for a high-priority curative autologous transplant
* Patients with rapidly progressive aggressive NHL unless in minimal disease state
* Active central nervous system (CNS) involvement with disease
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Patients who are human immunodeficiency virus (HIV) positive
* Cardiac ejection fraction < 40%
* Severe defects in pulmonary function testing (defects are currently categorized as mild, moderate and severe) as defined by the pulmonary consultant, or receiving supplementary continuous oxygen
* Total bilirubin > 2 x the upper limit of normal
* Serum glutamate pyruvate transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) 4 x the upper limit of normal
* Karnofsky score < 50
* Patients with poorly controlled hypertension
* Patients with renal failure are eligible, however patients with renal compromise (serum creatinine greater than 2.0) will likely have further compromise in renal function and may require hemodialysis (which may be permanent) due to the need to maintain adequate serum cyclosporine levels
* DONOR:

  * Identical twin
  * Age less than 12 years
  * Pregnancy
  * Infection with HIV
  * Inability to achieve adequate venous access
  * Known allergy to G-CSF
  * Current serious systemic illness

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-05; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Risk of graft rejection defined as the absence of detectable peripheral blood donor T cells with the addition of fludarabine phosphate | Up to day 56
Incidence of acute grade II/IV GVHD | Up to day 90 after the last DLI
Incidence of chronic GVHD | Up to 24 months

SECONDARY OUTCOMES:
Incidence of myelosuppression (ANC < 500/ul for > 2 days, platelets < 20,000/ul for > 2 days) after initial PBSC infusion | Up to day 56
Response of malignancy to DLI | Up to 24 months
Incidence of aplasia after DLI | Up to 24 months
Dose of CD3+ cells required to convert mixed to full lymphoid chimeras | Up to 24 months
Incidence of non-relapse mortality | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241